CLINICAL TRIAL: NCT00324402
Title: Plasma Brain Natriuretic Peptide Levels in Pregnancy
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2005008
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Cardiomyopathy; Pregnancy
Keywords: brain natriuretic peptide; pregnancy; biomarker
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy pregnant women, 18-40

SUMMARY:
To evaluate the maternal blood concentrations of brain natriuretic peptide (BNP) during the second and third trimesters of a normal pregnancy. We will attempt to define a normal range for pregnancy and any outliers that may serve as markers for abnormal cardiovascular physiology.

DETAILED DESCRIPTION:
The brain natriuretic peptide (BNP) is a useful marker for volume overload, increased filling pressures and stretching of the myocardium. The current literature contains limited and unreliable information regarding normal BNP values in pregnancy. After baseline echocardiogram to detect individuals with asymptomatic structural defects, the participants will submit to 3 blood draws during the second and third trimester and at delivery to determine normal pregnancy values.

ELIGIBILITY:
Inclusion Criteria:

* women age 18 to 40
* second trimester of pregnancy

Exclusion Criteria:

* known cardiac or valvular disease,
* atrial fibrillation or other arrhythmia,
* pulmonary hypertension,
* chronic hypertension,
* hypertensive disorders of pregnancy,
* morbid obesity (BMI > 40 kg/meter squared)
* history of sleep apnea
* multiple gestation
* known renal dysfunction
* medications known to affect cardiac function
* current or past abnormal echocardiogram

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women, 18-40
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-08; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Sorensen, DO, Study Chair — Oklahoma State University Center for Health Sciences; John M Beal, DO, Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma, United States